CLINICAL TRIAL: NCT01555424
Title: Bioavailability of Casein-bound Vitamin D From Fortified Cheese and Its Effects on the Well-being of the Institutionalized Elderly
Brief Title: Vitamin D Fortified Cheese and Well-being in the Institutionalized Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Reinhold Vieth, Dr., University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: M2327
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: The Focus is to Assess 25-hydroxyvitamin D Levels and Well-being
Keywords: 25-hydroxyvitamin D; Institutionalized seniors; SF-36 survey; Winter

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose (Active Comparator)
  Interventions: Dietary Supplement: High dose
- Reference dose (Active Comparator)
  Interventions: Dietary Supplement: Reference dose

INTERVENTIONS:
Dietary Supplement: High dose — This arm of the study receives a higher dose of the vitamin D fortified cheese (28,000IU/ 50g of cheddar cheese eaten once a week).
  Arms: High dose
Dietary Supplement: Reference dose — This arm of the study receives a lower dose of the vitamin D fortified cheese (200IU/ 50g of cheddar cheese eaten once a week).
  Arms: Reference dose

SUMMARY:
The investigators hypotheses is that the consumption of the investigators vitamin D fortified cheese will result in an increase in serum 25-hydroxy vitamin D levels in older institutionalized adults. Also, the consumption of the cheese with the higher amount of vitamin D will result in an improvement in wellbeing scores.

DETAILED DESCRIPTION:
The institute of medicine increased the dietary reference intakes of vitamin D for all of the age groups. The Recommended Daily Allowance (RDA) is now 800 IU for older adults over the age of 70, and the Tolerable Upper Level (UL) is 4000 IU daily. Canadians are known to have an inadequate vitamin D status, and older institutionalized adults are particularly susceptible to this. One strategy to correct this is to fortify more kinds of foods with vitamin D. We have already demonstrated that we can get vitamin D into cheddar cheese and it is as biologically available as vitamin D in the liquid supplement.

This new project aims to optimize the fortification process and deliver all of the vitamin D into cheddar cheese, and to measure its bioavailability and related changes in well-being during winter. We will assess the well being of the older institutionalized adults by administering the SF-36v2 health survey.

ELIGIBILITY:
Inclusion Criteria:

* Lactose intolerance
* Generally "Healthy", unless disease status deemed clinically significant and unable to participate by the attending physician.

Exclusion Criteria:

* Hypercalcemia/hypercalciuria
* Interfering medications
* Significant sun exposure in the months before and during the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The bioavailability of vitamin D from cheddar cheese fortified with vitamin D, in older institutionalized adults | 2 months
  We are adminstering 2 doses of vitamin D fortified cheese. One cheese contains a higher 28,000 IU/week dose that we expect to see health benefits with. The other cheese contains a 200IU/week dose that is similar to the current milk fortification practice in Canada (100IU per serving).

SECONDARY OUTCOMES:
A change in wellbeing scores using an SF-36 survey in the older institutionalized adults | 2 months
  We have previously shown that a group of adults showed an improvement in their wellbeing scores after the consumption of 28,000 IU/week of vitamin D during the winter months. Therefore, we will assess whether well-being changes in older institutionalized adults after the consumption of the vitamin D fortifed cheese, by using an SF-36 well-being survey.

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Vieth, PhD,FCACB, Principal Investigator — U of Toronto, Mount Sinai Hospital; Pierre Geoffroy, MD, Principal Investigator — Aurora Retirement Centre
Locations (1):
- Kingsway Arms- Aurora Retirement Centre, Aurora, Ontario, Canada

REFERENCES:
- [Background] Wagner D, Sidhom G, Whiting SJ, Rousseau D, Vieth R. The bioavailability of vitamin D from fortified cheeses and supplements is equivalent in adults. J Nutr. 2008 Jul;138(7):1365-71. doi: 10.1093/jn/138.7.1365. PMID 18567762
- [Background] Vieth R, Kimball S, Hu A, Walfish PG. Randomized comparison of the effects of the vitamin D3 adequate intake versus 100 mcg (4000 IU) per day on biochemical responses and the wellbeing of patients. Nutr J. 2004 Jul 19;3:8. doi: 10.1186/1475-2891-3-8. PMID 15260882